CLINICAL TRIAL: NCT04883073
Title: Impact on Quality of Life by Additional Use of the Digital Health Application "Endo-App" to Standard Therapy: Monocentric, Prospective, Randomised Trial (ELEA)
Brief Title: Impact on Quality of Life of "Endo-App" (ELEA)
Acronym: ELEA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Collaborators: Endo Health GmbH (Industry)
Responsible Party: Principal Investigator, Dr. med. Sebastian Daniel Schäfer, Head of Department of Gynecology, University Hospital Muenster
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ELEA
Record Dates: First submitted 2021-05-06; First posted 2021-05-12 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Endometriosis; Endometriosis-related Pain; Quality of Life
Keywords: endometriosis; quality of life; Endo-App; EHP-5; Endometriosis Health Profile; digital therapeutics
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Intervention Model Description: monocentric single side blinded randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endo App use (Experimental): use of Endo App during trial
  Interventions: Device: Use of Endo App
- control (No Intervention): no use of Endo App during trial

INTERVENTIONS:
Device: Use of Endo App — Use of Endo App
  Arms: Endo App use

SUMMARY:
monocentric randomized controlled trial enrolment of endometriosis patients from certified endometriosis centers. Randomization to control group (no Endo App use) vs intervention group (Endo App use) 12 weeks use / no use of Endo App. Evaluation of quality of life at onset, at 4, 8 and 12 weeks by using endometriosis health profile (EHP) 5 as a global index. Statistical analysis of global index at the end minus global index at onset between control and intervention group.

DETAILED DESCRIPTION:
randomized controlled trial enrolment of patients with diagnosed endometriosis 300 patients in total, 150 patients per group, randomization to control group (no Endo App use) vs intervention group (12 weeks Endo App use). The Endo App is a german language certified medical device which can be used to monitor the disease and gives support by providing complementary, multimodal interventions to standard therapy and is commercially available. Purpose of this study is the evaluation of quality of life at onset and then at 4, 8 and 12 weeks by using endometriosis health profile (EHP) 5 as a global index. The secondary endpoints of this study to evaluate are Fatigue symptoms (FSSsurvey), pain- specific self-efficacy (FESS), difficulty in everyday life due to pain (PDI) and emotional wellbeing (DASS- 21)

ELIGIBILITY:
Inclusion Criteria:

Legal capacity

* Living in Germany
* Adequate german language skills
* Female biological gender
* Ages eligible for study ≥ 18 years
* Medical Diagnosis of endometriosis

Diagnosis verification by following documents:

1. Operation Report
2. Histological finding
3. MRI finding
4. Other medical examination documents with endometriosis diagnosis (for example sonography, colonoscopy, cystoscopy)

Owning a smartphone and having an internet access

Willingness and capability of using the smartphone device and the Endo App

Motivation to regularly fill out the questionnaries

Owning an e-mail address for App registration

Absence of exlusion criteria

Exclusion Criteria:

* Absence of inclusion criteria
* Pregnancy existing at survey period
* Ongoing hormonal fertility treatment or planned treatment within the next 12 weeks (artificial insemination as part of in vitro fertilization, such as IVF or ICSI, hormone injections for fertility treatment)
* Ongoing or within the next 12 weeks planned rehabilitation or multimodal pain therapy
* Planned change in hormone therapy (change of active substance, new start or discontinuation of therapy) in the next 12 weeks or change in hormone therapy within the last 8 weeks before the start of the study
* Endometriosis surgery planned in the next 12 weeks or endometriosis surgery performed within the last 8 weeks prior to study start
* Previous or existing access to Endo app or current prescription

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2023-01-26 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
EHP 5 | 12 weeks
  Change in Endometriosis Health Profile 5 (minimum value: 0 points, maximum value: 100 points, higher scores mean a worse outcome)

SECONDARY OUTCOMES:
FSS survey | 12 weeks
  Change over course of study
FESS survey | 12 weeks
  Change over course of study
PDI survey | 12 weeks
  Change over course of study
DASS-21 survey | 12 weeks
  Change over course of study
EHP 5 | 4 weeks
  Change between 1st and 2nd survey
EHP 5 | 8 weeks
  Change between 1st and 3rd survey

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian D Schäfer, MD PhD, Principal Investigator — University Hospital Münster, Germany
Locations (1):
- University Hospital Münster Germany, Münster, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No